CLINICAL TRIAL: NCT00359034
Title: Fetal Aortic Pulsewave Velocity: A Novel Doppler Ultrasound Method of Measuring the Biophysical Properties of the Fetal Aorta
Status: Withdrawn | Type: Observational
Why Stopped: Could not resolve technical difficulties
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H06-70016
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: Doppler ultrasound; pulsewave velocity; intrauterine growth restriction; Fetal Pulsewave Velocity
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We are interested in determining if we can measure the blood flow in the descending aorta (large blood vessel in the abdomen) of healthy fetuses and fetuses with growth restriction. An increasing number of adult diseases (e.g. heart and blood vessel disease) are recognized as potentially associated with fetal growth and development.

Pulse wave velocity (PWV) is a measure of blood flow in blood vessels. This is routinely measured in adults, and has recently been studied in children. The purpose of our study is to see if we can develop a simple ultrasound method to measure the PWV in fetuses.

The purpose of this study is to see if we can consistently measure the blood flow patterns in the fetal descending aorta (large blood vessel in the abdomen) of 20 healthy fetuses and 20 growth restricted fetuses using standard ultrasound techniques.

DETAILED DESCRIPTION:
Prospective subjects will be recruited through:

1. Recruitment posters placed in the DAP department at BCWH. A contact number for the research nurse will be included on the recruitment poster for interested subjects to contact.
2. The antepartum inpatient unit at BCWH. Prospective subjects will be identified by the charge nurse as those patients satisfying the inclusion and exclusion criteria. Potential subjects will be asked by the charge nurse if they are interested in meeting a study investigator or research nurse for more information.
3. The same subject can participate twice in the study, once before 28 weeks and once after 28 weeks, as long as 3 weeks have passed between the study periods. All subjects participating before 28 weeks will be asked during the consent process if they are interested in participating a second time. Subjects in agreement will be contacted by the study nurse by phone to arrange a second appointment.

Study Procedure

Subject Involvement Measuring the PWV requires placing 3 electrocardiography (ECG) leads over the maternal abdomen in various positions to detect the fetal ECG signal. We have established that the fetal ECG signal can be detected as a small deflection in the maternal ECG tracing. The fetal ECG signal will allow us to correlate the blood flow wave form in the descending aorta to the fetal cardiac cycle. The onset of the blood flow waveform will be assessed at two points (A and B) along the descending aorta using standard pulsed Doppler ultrasound techniques. Point A will be the aortic isthmus and Point B will be at or beyond the level of the renal arteries. Measurements will be obtained in the following sequence: 1) time required for waveform to travel from Point A to Point B; 2) distance (mm) between Point A and Point B; 3) fetal heart rate using M-mode. The time it takes for the waveform to travel the measured distance between points A and B, will allow us to calculate the PWV in that portion of the fetal aorta. This sequence of measurements will be repeated three times in each fetus.

Subject Protocol

1. Subjects will be asked to drink 500 cc of water prior to arrival to appointment to ensure adequate hydration (which can affect amniotic fluid volume).
2. Subjects will be asked to void prior to entering study room.
3. Subjects will placed in the left lateral decubitus supine position
4. Subjects will rest for 15 minutes prior to the start of the ultrasound examination. At this time, consents will be reviewed again, and the demographic information recorded.
5. ECG electrodes will applied to the maternal abdomen
6. Fetal biometry, AFI and umbilical artery Dopplers will be performed (if not done within past 48 hours).
7. PWV will be determined at three times, within 10 minutes.

The demographic and pregnancy information collected will include:

1. maternal age
2. gestational age at the time of the study
3. obstetrical history (gravida, term, preterm, abortus, living)
4. maternal smoking history
5. amniotic fluid volume
6. estimated fetal weight and/or growth parameter percentiles

The following information will be collected and recorded during the study ultrasound:

1. time required to obtain the PWV measurement
2. the calculated PWV
3. maternal blood pressure and pulse
4. fetal presentation
5. fetal heart rate
6. presence or absence of fetal activity or breathing during the study
7. AFI and UA Doppler waveforms.

ELIGIBILITY:
Inclusion Criteria:

Study Group N:

Singleton pregnancy between 20 weeks 0 days and 36 weeks 0 days Normal obstetrical ultrasound in DAP at BCWH between 20-36 weeks GA

Study Group IUGR:

Singleton pregnancy between 20 weeks 0 days and 36 weeks 0 days Obstetrical ultrasound in DAP at BCWH between 20-36 weeks GA demonstrating IUGR (abdominal circumference AC <10%) and one of: a)oligohydramnios (amniotic fluid index (AFI) <5%) or b)abnormal umbilical artery (UA) Dopplers (absent or reversed end-diastolic flow)

Exclusion Criteria:

Study Group N:

Gestational age <20 weeks or ≥36 weeks Multiple pregnancy Any known or suspected fetal structural anomaly (including cardiac) Chromosomal abnormalities (on amniocentesis or CVS) Abnormalities in fetal growth (AC <10%; AC >90%) Abnormalities in amniotic fluid volume (AFI <5% or >95%) Maternal hypertensive disorder (during or prior to pregnancy) Illicit drug use during pregnancy (cocaine, heroin, methamphetamine) Maternal medical history of any chronic illness requiring medication (eg lupus, asthma, etc.) Abnormal maternal serum triple screen (AFP ≥2.5MoM, hCG >3.0 MoM)

Study Group IUGR:

Gestational age <20 weeks or ≥36 weeks Multiple pregnancy Any known or suspected fetal structural anomaly (including cardiac) Chromosomal abnormalities (on amniocentesis or CVS) Normal fetal growth with AC ≥10% Illicit drug use during pregnancy (cocaine, heroin, methamphetamine)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Singleton pregnancy between 20-36 weeks GA presenting at British Columbia Women's Hospital.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Pressey, MD, Principal Investigator — The University of British Columbia